CLINICAL TRIAL: NCT04406870
Title: Sirolimus in the Treatment for Propranolol-resistant Infantile Hepatic Hemangioendothelioma
Brief Title: Sirolimus in the Treatment for Infantile Hepatic Hemangioendothelioma(IEEH)
Acronym: PRL-SRL-IHHE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRL-SRL-IHHE
Record Dates: First submitted 2020-05-17; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Hemangioendothelioma of Liver
Keywords: propranolol-resistant; sirolimus; infantile hepatic hemangioendothelioma
MeSH Terms: interventions — temsirolimus; Sirolimus; Propranolol

STUDY DESIGN:
Intervention Model Description: Recruiting patients with IHHE who have no response to propranolol after 3 months. Then propranolol combined with sirolimus will be given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): patients with propranolol-resistant IHHE are given propranolol combined with sirolimus
  Interventions: Drug: Sirolimus Oral Product; Drug: propranolol

INTERVENTIONS:
Drug: Sirolimus Oral Product — Patients with IHHE wil be treated with propranolol (1 mg / kg , twice a day, after meals), and then evaluation will be performed after 3 months (changes of the tumor size measured by ultrasound examination, and changes of tumor volume measured by abdominal enhancement CT).It will be admitted into the group once the tumor volume shrinks <30%.Then propanolol combined with sirolimus will be given. Propranolol will be given at 1mg/kg,twice a day and sirolimus will be given at 0.8mg/m²(body surface area), twice a day. Recording and doing assessment of tumor size, adverse effects as well as complicated symptoms.
  Other Names: TORISEL; rapamycin
Drug: propranolol — Patients with IHHE wil be treated with propranolol (1 mg / kg , twice a day, after meals), and then evaluation will be performed after 3 months (changes of the tumor size measured by ultrasound examination, and changes of tumor volume measured by abdominal enhancement CT).It will be admitted into the group once the tumor volume shrinks <30%.Then propanolol combined with sirolimus will be given. Propranolol will be given at 1mg/kg,twice a day and sirolimus will be given at 0.8mg/m²(body surface area), twice a day. Recording and doing assessment of tumor size, adverse effects as well as complicated symptoms.
  Other Names: xin de an (chinese name means making me comfortable)

SUMMARY:
Infantile hepatic hemangioendothelioma (IHHE) is an infantile hemangioma involving the liver.Since 2008, propranolol has been used for the treatment of hemangioma, and some researchers have also started to report the use of propranolol for the treatment of infantile hepatic hemangioma in children. Sirolimus can be used in patients with vascular malformations such as hemangiomas. IHHE is also an infantile hemangioma involving the liver,thus sirolimus may paly the role in treatment of IHHE.The clinical trial explores the efficacy of sequential treatment of sirolimus to refractory IHHE patients resistant with propranolol, to improve the therapeutic effect, reduce the side effects of traditional treatment methods (hormones, interferon), and reduce the number of operations and interventions and to provide a clinical basis for the application of the new therapeutics model of IHHE of "propranolol + sequential sirolimus treatment".

DETAILED DESCRIPTION:
According to the World Health Organization(WHO) classification of digestive system tumors in the fourth edition in 2010, infantile hepatic hemangioendothelioma (IHHE) is an infantile hemangioma involving the liver. It is a benign tumor, which can be subgrouped into focal, multifocal, and diffusing in children, as well as combining vascular malformations of the skin, brain, digestive tract and other organs.Since 2008, propranolol has been used for the treatment of hemangioma, and some researchers have also started to report the use of propranolol for the treatment of infantile hepatic hemangioma in children.And more and more clinicians unanimously recommend propranolol as first-line medication for the treatment of IHHE.However, there are few solutions to propranolol-resistant IHHE. Sirolimus is a serine/threonine kinase which plays a pivotal role in cell mortality, angiogenesis and cell growth. Sirolimus can be used in patients with vascular malformations such as hemangiomas. Children with vascular malformations received 0.1mg/kg of sirolimus orally every day and maintained the blood concentration at 8-15ng/ml. The lesions gradually disappear with time going on. Therefore, sirolimus can be used as a second-line medicine for refractory hemangioma and vascular malformation.Interestingly, the investigator's previous study which is retrospective analysis of 30 patients has indicated the effective rate of propranolol alone in treating infantile hepatic endothelial tumor (IHHE) was 57.7%, while that of sequential treatment combined with sirolimus was 84.6%.So, this clinical trial is going to explore the efficacy of sequential treatment of sirolimus to refractory IHHE patients resistant with propranolol,to improve the therapeutic effect,furtherly, reduce the side effects of traditional treatment methods (hormones, interferon), as well as the number of operations and interventions and to provide a clinical guide for the novel therapeutics model of propranolol combined with sirolimus for sequential treatment of infantile hepatic hemangioendothelioma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed as IHHE
* Age between 1 month and 36 months
* Receiving propranolol for 3 months but the tumor size shrinks <30%
* With written informed consent

Exclusion Criteria:

* Confirmed as hepatoblastoma
* Have accepted surgical resection
* Clinical data missing
* Patients with Kasabach-Merritt phenomenon
* Receiving propranolol for 3 months and the tumor size shrinks >30%

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of tumor size | 1 month
  measuring the tumor size by ultrasound

SECONDARY OUTCOMES:
Change of PIVKA-II | 1 month
  Using PIVKA-II assay kit (ARCHITECT I2000SR REFURB, Abbott, America).
Change of alpha-1 fetoprotein (AFP) | 1 month
  Using the AFP assay kit (ARCHITECT AFP, Abbott, America).

CONTACTS AND LOCATIONS:
Overall Officials: Song Gu, Doctor, Study Chair — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Requena L, Kutzner H. Hemangioendothelioma. Semin Diagn Pathol. 2013 Feb;30(1):29-44. doi: 10.1053/j.semdp.2012.01.003. PMID 23327728
- [Background] Chatmethakul T, Bhat R, Alkaabi M, Siddiqui A, Peevy K, Zayek M. Infantile Hepatic Hemangioendothelioma: An Uncommon Cause of Persistent Pulmonary Hypertension in a Newborn Infant. AJP Rep. 2016 Jul;6(3):e260-3. doi: 10.1055/s-0036-1585578. PMID 27468364
- [Background] Chen CC, Kong MS, Yang CP, Hung IJ. Hepatic hemangioendothelioma in children: analysis of thirteen cases. Acta Paediatr Taiwan. 2003 Jan-Feb;44(1):8-13. PMID 12800377
- [Background] Mehrabi A, Kashfi A, Schemmer P, Sauer P, Encke J, Fonouni H, Friess H, Weitz J, Schmidt J, Buchler MW, Kraus TW. Surgical treatment of primary hepatic epithelioid hemangioendothelioma. Transplantation. 2005 Sep 27;80(1 Suppl):S109-12. doi: 10.1097/01.tp.0000186904.15029.4a. PMID 16286886
- [Background] Maaloul I, Aloulou H, Hentati Y, Kamoun T, Mnif Z, Hachicha M. Infantile hepatic hemangioendothelioma successfully treated by low dose of propranolol. Presse Med. 2017 Apr;46(4):454-456. doi: 10.1016/j.lpm.2017.01.010. Epub 2017 Mar 15. No abstract available. PMID 28318668
- [Background] Chaturvedi K, Steinberg JS, Snyder CS. Cost-effectiveness of treating infantile haemangioma with propranolol in an outpatient setting. Cardiol Young. 2018 Oct;28(10):1105-1108. doi: 10.1017/S1047951118000987. Epub 2018 Jul 26. PMID 30047346
- [Background] Avagyan S, Klein M, Kerkar N, Demattia A, Blei F, Lee S, Rosenberg HK, Arnon R. Propranolol as a first-line treatment for diffuse infantile hepatic hemangioendothelioma. J Pediatr Gastroenterol Nutr. 2013 Mar;56(3):e17-20. doi: 10.1097/MPG.0b013e31824e50b7. No abstract available. PMID 22331019
- [Background] Ozdemir ZC, Duzenli Kar Y, Sohret NC, Kebapci M, Bor O. Beta blocker and steroid therapy in the treatment of infantile hepatic hemangioendothelioma. Drug Discov Ther. 2017 Jul 31;11(3):161-164. doi: 10.5582/ddt.2017.01025. Epub 2017 Jul 25. PMID 28652510